CLINICAL TRIAL: NCT00189878
Title: Multi-centre Prospective Randomised Double-blind Placebo-controlled Study of Methotrexate in the Treatment of Chronic Idiopathic Urticaria
Brief Title: A Study of the Use of Methotrexate in the Treatment of Chronic Idiopathic Urticaria
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: unable to recruit
Sponsor: Barnsley Hospital (Other)
Responsible Party: Jeffrey Bailey, Research and Development, Barnsley Hospital NHS Foundation Trust
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MREC/03/4/003; MF 8000/12375
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Urticaria
Keywords: chronic idiopathic urticaria; methotrexate
MeSH Terms: conditions — Urticaria; Chronic Urticaria | interventions — Methotrexate; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 methotrexate (Active Comparator): patient to receive methotrexate
  Interventions: Drug: Methotrexate (drug)
- 2 Placebo (Placebo Comparator): given placebo capsules
  Interventions: Drug: placebo capsules

INTERVENTIONS:
Drug: Methotrexate (drug) — Methotrexate 10 to 15 mg weekly for 8 weeks
  Arms: 1 methotrexate
Drug: placebo capsules — 4-6 placebo capsules - identical to capsules containing methotrexate
  Arms: 2 Placebo

SUMMARY:
The purpose of this study is to determine whether methotrexate produces significant improvement in chronic idiopathic urticaria, compared with placebo

DETAILED DESCRIPTION:
Chronic idiopathic urticaria is thought to affect approximately 0.1% of the population. It can be very disabling and difficult to treat. Antihistamines are the only drugs licensed for treatment of urticaria, however there is a group of severely affected patients with chronic idiopathic urticaria who fail to respond. Previous trials have shown ciclosporin to be beneficial, and small studies support the use of intravenous immunoglobulins and plasmapheresis. However, not only are these options expensive, but since chronic idiopathic urticaria may persist for years, their prolonged use may be limited by adverse effects. We have previously published a report of 2 patients who responded to methotrexate, and wish to properly evaluate the efficacy of methotrexate in the treatment of CIU.

In the first part of the study patients will be given either placebo or methotrexate for 8 weeks and in the second part of the study, non-responders will be offered open labelled methotrexate for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* severe unremitting chronic idiopathic urticaria
* disease resistant to treatment with antihistamines
* aged 18 years or more

Exclusion Criteria:

* predominant physical urticaria
* urticarial vasculitis
* any contraindication to the use of methotrexate, eg. pregnancy / breast feeding, women wanting to conceive or man wanting to father a child within 12 months of entry, use of drugs which interact, underlying medical conditions
* use of immunosuppressant within 4 weeks of entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2003-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
A positive response to treatment (a reduction to <25% of baseline urticaria activity scores) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ruth A Sabroe, FRCP, MD, Principal Investigator — Barnsley Hospital NHS Foundation Trust